CLINICAL TRIAL: NCT01294696
Title: Survey of Osteoarthritis Real World Therapies (SORT)
Brief Title: Survey of Osteoarthritis Real World Therapies (MK-0663-140)
Acronym: SORT
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: 0663-140
Record Dates: First submitted 2010-12-22; First posted 2011-02-11 (Estimated); Results first posted 2014-03-04 (Estimated); Last update posted 2024-08-29 (Actual); Status verified 2022-02

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Standard of care
MeSH Terms: conditions — Osteoarthritis | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Enrolled Participants: All participants will be treated according to standard medical guidelines or usual clinical practice standards of the investigating physician.
  Interventions: Drug: Standard of care for treatment of osteoarthritis (OA) of knee(s)

INTERVENTIONS:
Drug: Standard of care for treatment of osteoarthritis (OA) of knee(s) — All participants will be treated according to standard medical guidelines or usual clinical practice standards of the investigating physician.

SUMMARY:
This was a study to estimate the proportion of participants with osteoarthritis of the knee(s) who were treated with oral or topical analgesics for their symptoms, who did and did not report adequate pain relief at Baseline and to characterize their pain level over a 12-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary osteoarthritis of the knee(s)
* Presently receiving prescribed oral or topical analgesics for a minimum duration of two weeks prior to enrollment

Exclusion Criteria:

* Arthritis other than primary osteoarthritis
* Treatment with disease-modifying antirheumatic drugs (DMARDS), methotrexate or biologics
* Subtotal or total joint replacement in the affected knee
* Chronic severe pain of other causes that in the opinion of the investigator may require long-term analgesia or confound the present study
* Currently enrolled in a clinical trial or who have participated in a clinical trial within the past 30 days

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who are presently receiving prescribed oral or topical analgesics which commenced at least two weeks prior to enrollment
Sampling Method: Non-Probability Sample
Enrollment: 1261 (Actual)
Dates: Start 2010-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

REFERENCES:
- [Result] Conaghan PG, Peloso PM, Everett SV, Rajagopalan S, Black CM, Mavros P, Arden NK, Phillips CJ, Rannou F, van de Laar MA, Moore RA, Taylor SD. Inadequate pain relief and large functional loss among patients with knee osteoarthritis: evidence from a prospective multinational longitudinal study of osteoarthritis real-world therapies. Rheumatology (Oxford). 2015 Feb;54(2):270-7. doi: 10.1093/rheumatology/keu332. Epub 2014 Aug 23. PMID 25150513

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 54 trial centers: 18 in France; 4 in Italy; 5 in The Netherlands; 5 in Portugal; and 9 in the United Kingdom.
Groups:
- All Enrolled Participants: The population consisted of all enrolled participants with adequate and inadequate pain relief.
Period: Overall Study
Arm/Group | All Enrolled Participants
Started | 1261
Completed | 1187
Not Completed | 74
Not completed — Screening failures | 7
Not completed — Protocol Violation | 8
Not completed — Missing BPI Response | 7
Not completed — Site closure | 52

BASELINE CHARACTERISTICS:
Groups:
- Participants With Adequate Pain Relief: Adequate pain relief was defined as an average pain score of <=4 on the Brief Pain Inventory (BPI). Baseline characteristics are only reported for participants with data available at baseline.
- Participants With Inadequate Pain Relief: Inadequate pain relief was defined as an average pain score of >4 on the BPI. Baseline characteristics are only reported for participants with data available at baseline.
- Total: Total of all reporting groups
Arm/Group | Participants With Adequate Pain Relief | Participants With Inadequate Pain Relief | Total
Number analyzed (Participants) | 548 | 639 | 1187
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.6 (9.03) | 68.0 (9.76) | 67.8 (9.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 329 | 479 | 808
  Male | 219 | 160 | 379

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Reported Adequate vs. Inadequate Pain Relief at Baseline
Description: Participant pain at baseline was recorded using the Brief Pain Inventory (BPI). The BPI is an inventory of subject-reported questions, where for each pain severity item the response scale is 0 = No Pain and 10 = Worst Pain You Can Imagine. The questions refer to pain due to osteoarthritis in the affected knee in the last week: at its worst, at its least, on the average, and right now. Adequate pain control was defined as a score of <=4 on question 5 of the BPI. Inadequate pain control was defined as a score >4 on question 5 of the BPI. Question 5 of the BPI asked participants to rate their pain by circling the number that best describes their pain on the average scale from 0 to 10 (with 0=no pain and 10=worst pain imaginable).
Time Frame: Baseline (Day 1)
Population: The population consisted of all participants for which a BPI value was available at baseline.
Measure: Number; unit: Percentage of Participants
Groups:
- All Enrolled Participants: All enrolled participants that were treated with the local standard of care for osteoarthritis of the knee.
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 1187
Percentage of Participants
  Adequate Pain Relief | 46.2
  Inadequate Pain Relief | 53.8

2. Primary Outcome: Percentage of Participants Who Reported Adequate vs. Inadequate Pain Relief at Month 12
Description: Participant pain at baseline was recorded using the Brief Pain Inventory (BPI). The BPI is an inventory of subject-reported questions, where for each pain severity item the response scale is 0 = No Pain and 10 = Worst Pain You Can Imagine. The questions refer to pain in the last week: at its worst, at its least, on the average, and right now. Adequate pain control was defined as a score of <=4 on question 5 of the BPI. Inadequate pain control was defined as a score >4 on question 5 of the BPI. Question 5 of the BPI asked participants to rate their pain by circling the number that best describes their pain on the average scale from 0 to 10 (with 0=no pain and 10=worst pain imaginable).
Time Frame: Month 12
Population: The population consisted of all participants for which a BPI value was avaialble at Month 12.
Measure: Number; unit: Percentage of Participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 1074
Percentage of Participants
  Adequate Pain Relief | 47.3
  Inadequate Pain Relief | 52.7

3. Secondary Outcome: Percentage of Participants Who Reported Adequate Relief From Joint Stiffness or Limitation in Physical Function at Baseline (Day 1)
Description: Joint stiffness or limitation in physical function was evaluated using the Western Ontario and McMasters Universities (WOMAC) visual analog (VA)3.0 Index. The WOMAC VA 3.0 is a self-administered, tri-dimensional, disease-specific health status measure. It probes clinically important, subject-relevant symptoms in the areas of pain, joint stiffness and physical function in subjects with osteoarthritis of the knee. The index consists of 24 questions (5 pain, 2 stiffness and 17 physical function) and uses a VA scale of 0-500 mm for pain, 0-200 mm for stiffness, and 0-1700 for physical limitation with higher scores indicating poorer outcomes. Adequate pain was defined as participants reporting less than 4 on the BPI average pain scale.
Time Frame: Baseline (Day 1)
Population: The population consisted of all participants for which WOMAC VA 3.0 data for joint stiffness and limiation in physical function were available at Baseline.
Measure: Number; unit: Percentage of Participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 1097
Percentage of Participants | 43.4

4. Secondary Outcome: Percentage of Participants Who Reported Adequate Relief From Joint Stiffness or Limitation in Physical Function at Month 1
Description: Joint stiffness or limitation in physical function was evaluated using the Western Ontario McMaster Osteoarthritis (WOMAC) visual analog (VA)3.0 Index. The WOMAC VA 3.0 is a self-administered, tri-dimensional, disease-specific health status measure. It probes clinically important, subject-relevant symptoms in the areas of pain, joint stiffness and physical function in subjects with osteoarthritis of the knee. The index consists of 24 questions (5 pain, 2 stiffness and 17 physical function) and uses a VA scale of 0-500 mm for pain, 0-200 mm for stiffness, and 0-1700 for physical limitation with higher scores indicating poorer outcomes. Adequate pain was defined as participants reporting less than 4 on the BPI average pain scale.
Time Frame: Month 1
Population: The population consisted of all participants for which a WOMAC VA 3.0 measurement was available at Month 1.
Measure: Number; unit: Percentage of Participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 1026
Percentage of Participants | 44.8

5. Secondary Outcome: Percentage of Participants Who Reported Adequate Relief From Joint Stiffness or Limitation in Physical Function at Month 3
Description: as for outcome 3
Time Frame: Month 3
Population: The population consisted of all participants for which WOMAC VA 3.0 data were available at Month 3.
Measure: Number; unit: Percentage of Participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 1013
Percentage of Participants | 44.7

6. Secondary Outcome: Percentage of Participants Who Reported Adequate Relief From Joint Stiffness or Limitation in Physical Function at Month 6
Description: as for outcome 3
Time Frame: Month 6
Population: The population consisted of all participants for which WOMAC VA 3.0 data were available at Month 6.
Measure: Number; unit: Percentage of Participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 1070
Percentage of Participants | 45.3

7. Secondary Outcome: Percentage of Participants Who Reported Adequate Relief From Joint Stiffness or Limitation in Physical Function at Month 9
Description: as for outcome 3
Time Frame: Month 9
Population: The population consistated of all participants for which WOMAC VA 3.0 data were available at Month 9.
Measure: Number; unit: Percentage of Participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 1039
Percentage of Participants | 48.6

8. Secondary Outcome: Percentage of Participants Who Reported Adequate Relief From Joint Stiffness or Limitation in Physical Function at Month 12
Description: as for outcome 3
Time Frame: Month 12
Population: The population consisted of all participants for which WOMAC VA 3.0 data was available at Month 12.
Measure: Number; unit: Percentage of Participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 1058
Percentage of Participants | 49.6

ADVERSE EVENTS:
Time Frame: Up to Month 12
Groups:
- Participants With Adequate Pain Relief: Adequate pain relief was fedined as an average pain score of <=4 on the Brief Pain Inventory (BPI).
Arm/Group | Participants With Adequate Pain Relief | Participants With Inadequate Pain Relief
Serious Adverse Events (participants affected / at risk) | 11/548 | 25/639
Other Adverse Events (participants affected / at risk) | 0/548 | 0/639
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Adequate Pain Relief (N=548) | Participants With Inadequate Pain Relief (N=639)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina Unstable (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (2)
Abdominal Distention (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Localized Infection (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Periumbilical Abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Burns Third Degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's Disease (Nervous system disorders) | 0 (0) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1) | 0 (0)
Calculus Bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral Sclerosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.